CLINICAL TRIAL: NCT03850418
Title: Azacitidine and Chimerism in MDS or AML Patients After Allogeneic Stem Cell Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, Principal Investigator, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12592
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Myeloid Malignancy
MeSH Terms: interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AZA (Experimental): azacitidine
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: azacitidine — azacitidine 32mg/m2 x 5 days every 28 days for minimum of 4 cycles if tolerated

SUMMARY:
Previous studies provide a rationale for administration of AZA after allo SCT for decreasing chimerism. The investigators hypothesize that azacitidine can be well tolerated after SCT and help decrease rate of decreasing donor chimerism and hence decrease relapse without increasing GVHD

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AML/MDS/MPN, CMML post Allogeneic SCT who experience any drop in total or myeloid chimerism any time after day 30, or their day 30 or day100 myeloid donor chimerism is below 98% without concurrent hematologic relapse (that is, patients with <5% bone marrow blasts as obtained at that time point) will be offered treatment with azacitidine
2. >=30 -180 days post SCT and patients must have ANC> 1000, PLT > 50,000
3. Age 18-75 years old
4. Performance score of at least 70% by Karnofsky
5. Adequate kidney and liver function as demonstrated by:

   1. Creatinine clearance should be >60 ml/min
   2. Total Bilirubin <1.5, ALT/AST/Alk Phos < 2.5 x normal. No evidence of chronic active hepatitis or cirrhosis.
6. Negative Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use an effective contraceptive measure while on study.
7. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.
8. Patients must be off any prior chemotherapy, radiotherapy, or other investigational therapy within 2 weeks prior to start treatment

Exclusion Criteria:

1. Positive for HIV, HBsAg, HCV or other viral hepatitis or cirrhosis from any cause
2. Active or prior CNS leukemia, unless in complete remission for at least 2 months.
3. History of serious chronic mental disorder or drug-abuse accompanied by documented problems of compliance with therapeutic programs.
4. Uncontrolled infection
5. Grade III, IV graft versus host disease (GVHD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The rate of increase or stable donor chimerism | one year
  To determine the rate of increase or stable donor chimerism when using low dose azacitidine post allogenic stem cell transplant (SCT) in patients with acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML) and myeloproliferative neoplasms (MPN) with documented low or decreasing donor chimerism

CONTACTS AND LOCATIONS:
Locations (1):
- Henry ford hospital, Detroit, Michigan, United States